CLINICAL TRIAL: NCT04702555
Title: Analgesic Efficacy of Orally Administered VTS-K (Liquid Oral Ketamine Taken Simultaneously With VTS-Aspirin) for Pain Management of Adult ED Patients Presenting to the ED With Acute Musculoskeletal Pain
Brief Title: Analgesic Efficacy of Orally Administered VTS-K for Pain Management
Status: Completed | Type: Observational
Sponsor: Antonios Likourezos (Other)
Responsible Party: Sponsor-Investigator, Antonios Likourezos, Research Manager, Maimonides Medical Center
Organization: Maimonides Medical Center (Other)
Other Study IDs: 2020-10-17-MMC
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Pain, Acute
Keywords: Pain; Pain Management; Ketamine; Emergency Medicine
MeSH Terms: conditions — Acute Pain; Pain; Agnosia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Vitalis Pharmaceuticals (VTS)-Aspirin and Ketamine: An oral combination drug of VTS-Aspirin and ketamine (VTS-K) would facilitate the shift from IV opioids to a non-IV therapy for patients presenting to the ED with acute MSK pain. This formulation has a potential to provide effective analgesia in the ED with reduced side effects. VTS-K's proprietary oral formulation of established, safe, and well-understood APIs, makes it uniquely appropriate for use in the ED. VTS-K is administered orally, which is suitable for resource-poor environments in which the healthcare setting may be inadequate as well as suitable to improve the throughput of ED Patients by reducing their length of stay. This is especially pertinent given the alternative of IV opioids for pain management of acute MSK pain, which requires both clinical monitoring and equipment, whereas VTS-K promotes weaning off opioids, alleviating the resource consumption.
  Interventions: Drug: VTS-K

INTERVENTIONS:
Drug: VTS-K — An oral combination drug of VTS-Aspirin and ketamine (VTS-K)

SUMMARY:
A combination of ketamine and aspirin for the treatment of acute MSK pain in the ED would confer multimodal analgesia, with the contributions of aspirin and ketamine to an opioid sparing effect. Research on this multimodal approach is sparse, but the minimal empirical evidence supports a clinical benefit to patients in a post orthopedic surgery setting, both in short term and long term.

Vitalis Pharmaceuticals (New York, NY) has developed a proprietary formulation of aspirin, VTS-Aspirin, that may deliver faster and stronger pain reduction than traditional aspirin. Preliminary research indicates that combinations of VTS-Aspirin with analgesics may confer greater benefit in pain management than some current standards of care (26).

An oral combination drug of VTS-Aspirin and ketamine (VTS-K) would facilitate the shift from IV opioids to a non-IV therapy for patients presenting to the ED with acute MSK pain. This formulation has a potential to provide effective analgesia in the ED with reduced side effects. VTS-K's proprietary oral formulation of established, safe, and well-understood APIs, makes it uniquely appropriate for use in the ED. VTS-K is administered orally, which is suitable for resource-poor environments in which the healthcare setting may be inadequate as well as suitable to improve the throughput of ED Patients by reducing their length of stay. This is especially pertinent given the alternative of IV opioids for pain management of acute MSK pain, which requires both clinical monitoring and equipment, whereas VTS-K promotes weaning off opioids, alleviating the resource consumption.

DETAILED DESCRIPTION:
STUDY OBJECTIVES

To evaluate analgesic efficacy of orally administered VTS-K (liquid oral ketamine taken simultaneously with VTS-Aspirin and oral ketamine (in a liquid form)) for pain management of adult ED patients presenting to the ED with acute musculoskeletal pain

HYPOTHESIS

In our pilot study we hypothesize that the VTS-K combination will result in analgesia with a change in pain score at least of 1.3 points on NRS. The primary outcome of this trial is the reduction in participant's pain scores at 60 minutes post medication administration.

STUDY DESIGN

Subjects: Patients 18 years of age and older presenting to the ED with acute musculoskeletal painful conditions (traumatic and non-traumatic) with a an initial pain score of 5 or more on a standard 11- point (0 to 10) numeric rating scale and requiring oral analgesia as determined by the treating attending physician. Patients' screening and enrollment will be performed by study investigators and research assistants. All patients will be enrolled at various times of the day when study investigators will be available for patient enrollment and an ED pharmacist will be available for medication preparation

Eligibility Criteria: Patients 18 years of age and older presenting to the ED with acute musculoskeletal painful conditions (traumatic and non-traumatic) with an initial pain score of 5 on a standard 11- point (0 to 10) numeric rating scale. Patients will have to be awake, alert, and oriented to person, place, and time, and will be able to demonstrate understanding of the informed consent process and content. Patients also will have to demonstrate ability to verbalize the nature of any adverse effects they might experience as well as to express their pain severity by using the NRS.

Exclusion Criteria: Patients with altered mental status, allergy to aspirin and ketamine, pregnant patients, unstable vital signs (systolic blood pressure <90 or>180 mm Hg, pulse rate <50 or >150 beats/min, and respiration rate <10 or >30 breaths/min), inability to provide consent, consumption of Aspirin or NSAID's within 6 hours of arrival to the ED, active PUD, history of GI Hemorrhage, history of renal and hepatic insufficiency, past medical history of alcohol or drug abuse, or schizophrenia.

Design: This is a prospective observational pilot trail evaluating analgesic efficacy and safety of VTS-K in adult patients presenting to the ED of Maimonides Medical Center with acute musculoskeletal painful conditions. Upon meeting the eligibility criteria, patients will be offered to participate in the study.

Data Collection Procedures: Each patient will be approached by a study investigator for acquisition of written informed consent and Health Insurance Portability and Accountability Act authorization after being evaluated by the treating emergency physician and determined to meet study eligibility criteria. When English will not be the participant's primary language, a language- appropriate consent form will be used and non-investigator, hospital-employed, trained interpreters or licensed telephone interpreter will assist in acquisition of informed consent. Baseline pain score will be determined with an 11-point numeric rating scale (0 to 10), described to the patient as "no pain" being 0 and "the worst pain imaginable" being 10. A study investigator will record the patient's body weight and baseline vital signs.

The on-duty ED pharmacist will prepare an oral dose of ketamine by using a formulary for parenteral use. The oral dosing regimen of ketamine is 0.5 mg/kg that will be placed in the syringe or a medication cup. The research associate will deliver both medications (VTS-Aspirin and Oral Ketamine) to the patient. Study investigators will record pain scores and adverse effects at 15, 30, 60, and 90 minutes. If patients reported a pain numeric rating scale score of 5 or greater and requested additional pain relief, an oral immediate release morphine tablet of 7.5 mg will be given

All data will be recorded on data collection sheets, including patients' sex, demographics, medical history, and vital signs, and entered into SPSS (version 24.0; IBM Corp) by the research manager. Confirmation of written consent acquisition for all participants, and statistical analyses will be conducted by the statistician, who will work independently of any data collection.

Patients will be closely monitored for adverse effects during the entire study period (up to 90 minutes) by study investigators. Common adverse effects that are associated with oral ketamine are felling of unreality, dizziness, nausea, vomiting, and sedation. Common adverse effects are associated with VTS-Aspirin are nausea, dyspepsia, epigastric discomfort.

ELIGIBILITY:
Inclusion Criteria:

* 18 years+
* presenting to Maimonides Medical Center ED
* acute musculoskeletal painful conditions (traumatic and non-traumatic) with an initial pain score of 5 on a standard 11- point (0 to 10) numeric rating scale
* be awake, alert, and oriented to person, place, and time,
* demonstrate understanding of the informed consent process and content.
* have to demonstrate ability to verbalize the nature of any adverse effects they might experience as well as to express their pain severity by using the NRS.

Exclusion Criteria:

* Patients with altered mental status
* allergy to aspirin and ketamine
* pregnant patients
* unstable vital signs (systolic blood pressure <90 or>180 mm Hg
* pulse rate <50 or >150 beats/min
* respiration rate <10 or >30 breaths/min)
* inability to provide consent
* consumption of Aspirin or NSAID's within 6 hours of arrival to the ED
* active PUD
* history of GI Hemorrhage
* history of renal and hepatic insufficiency
* past medical history of alcohol or drug abuse
* schizophrenia.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age and older presenting to the ED with acute musculoskeletal painful conditions (traumatic and non-traumatic) with a an initial pain score of 5 or more on a standard 11- point (0 to 10) numeric rating scale and requiring oral analgesia as determined by the treating attending physician. Patients' screening and enrollment will be performed by study investigators and research assistants. All patients will be enrolled at various times of the day when study investigators will be available for patient enrollment and an ED pharmacist will be available for medication preparation
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2021-01-08 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
The analgesic efficacy of orally administered VTS-K (liquid oral ketamine taken simultaneously with VTS-Aspirin and oral ketamine (in a liquid form)) for pain management of adult ED patients presenting to the ED with acute musculoskeletal pain | 30 minutes
  To assess whether VTS-K is effective in reducing acute MSK pain in ED patients using a 11 Point Likert Scale with 0 being no pain, 5 being moderate pain, and 10 being severe pain.

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Motov, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davis A, Fassassi C, Dove D, Drapkin J, Likourezos A, Gohel A, Favale P, Hossain R, Butt M, Gerges L, Motov S. Analgesic Efficacy of Oral Aspirin/Ketamine Combination for Management of Acute Musculoskeletal Pain in the Emergency Department - A Proof of Concept Pilot Study. J Emerg Med. 2022 Jun;62(6):750-759. doi: 10.1016/j.jemermed.2022.01.029. Epub 2022 May 24. PMID 35624056

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-19): https://cdn.clinicaltrials.gov/large-docs/55/NCT04702555/Prot_SAP_000.pdf